CLINICAL TRIAL: NCT05555927
Title: Adjunctive Duration-doubled Transcranial Direct Current Stimulation (tDCS) for the Treatment of Depressive Patients With Suicidal Ideation: Study Protocol for a Double-blind, Randomized, Sham-controlled Trial
Brief Title: Adjunctive Duration-doubled tDCS for the Treatment of Depressive Patients With Suicidal Ideation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Yiming Chen, Principal Investigator, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-SMHCYJXYS-06
Record Dates: First submitted 2022-09-14; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Experimental): tDCS devices (Neuroelectrics, Starstim 8, USA) are used. The anode and cathode electrodes are inserted in saline-soaked sponges with diameter of 3.2cm and then positioned over the left and right dorsolateral prefrontal cortex (DLPFC) using specific headgear. Each session uses a 2mA current and lasts 60 minutes. Ten sessions are daily performed.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- sham tDCS (Sham Comparator): The anode and cathode electrodes are inserted in saline-soaked sponges with diameter of 3.2cm and then positioned over the left and right dorsolateral prefrontal cortex (DLPFC) using specific headgear. Each session uses a 2mA current and lasts 60 minutes. Ten sessions are daily performed. For sham, the current rapidly ramp up to 2mA over the first 30s and rapidly ramped down to 0mA over the next 30s automatically to allow participants to feel typical initial sensations of active tDCS.
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation is an non-invasive brain stimulation that is proposed as a possible interventional tool for major depressive disorder. tDCS device that this study used is from Neuroelectrics, Starstim 8, USA.

SUMMARY:
In this double-blinded, randomized, sham-controlled trial, the investigators aim to determine the acute effectiveness of duration-doubled tDCS on suicidal ideation in patients with MDD. In addition to the their usual treatment, participants will be randomly assigned to receive either 10 weekday sessions of active (2 mA) or sham tDCS as an adjunctive treatment, with the anode over the left DLPFC and the cathode over the right DLPFC. The investigators will regularly assess suicidal ideation, depression severity and functional impact using the BSI, HAMD-17, MADRS, ODQ, YMRS, ASRM, CGI and SDS throughout the trial. The investigators will assess cognitive changes using WCST and SCWT. The investigators will also regularly assess treatment-related side effects using validated scales.

DETAILED DESCRIPTION:
Backgroud: During the last decade, the problem of suicide has become increasingly common in individuals with depression. Transcranial direct current stimulation (tDCS) is an effective treatment for major depressive disorder (MDD) with 2 milliamperes (mA) for at least thirty minutes per day for two weeks.

Aims: To investigate the efficacy of daily duration-doubled performed tDCS as an adjunctive intervention for rapidly improving suicidal ideation and depression in MDD patients with antidepressants.

Methods and design: In this double-blind, randomized, sham-controlled study, 76 MDD patients with suicidal ideation will be randomly assigned to either active (n=38) or sham (n=38) tDCS group. The anode and the cathode are placed over the scalp areas corresponding to the left and the right dorsolateral prefrontal cortex (DLPFC), respectively, and the stimulation lasts for 60 minutes. The primary outcome, severity of suicidal ideation, is measured by the Beck Scale for Suicide Ideation (BSI). The 17-item Hamilton Depression Rating Scale (HAMD-17) and Montgomery-Asberg Depression Rating Scale (MADRS) are utilized to assess the severity of depression. The Wisconsin Card Sorting Test (WCST) and Stroop Color-Word Test (SCWT) are adopted to assess executive function. Blood biomarkers are collected at baseline, after the 5th intervention and at the end of 10th intervention to calculate white blood cell (WBC), C-reactive protein (CRP), neutrophils, lymphocytes, monocytes, platelets and MDD related cytokines such as nerve growth factor (NGF), brain-derived (BDNF), glial-cell line derived neurotrophic factor (GDNF), the interleukins (IL), tumor necrosis factor-alpha (TNF-alpha), and its soluble receptors sTNFr1 and sTNFr2. The investigators hypothesis that, in contrast to the sham group, the active tDCS group may show a superiority in BSI, HAMD-17, MADRS score reduction after 5 and 10 sessions. Moreover, the investigators will evaluate associations of the improvement of suicidal ideation with the variation of WBC, CRP, neutrophils, lymphocytes, monocytes, platelets, neutrophil-to-lymphocyte ratio (NLR), monocyte-to-lymphocyte ratio (MLR), and platelet-to-lymphocyte ratio (PLR) count.

Conclusions: This study suggest that the adjunctive duration-doubled tDCS might be a novel method to rapidly reduce suicidal ideation and improve depressive symptom. And the variation of peripheral markers could be potential biomarkers of suicide risk and severity of MDD.

ELIGIBILITY:
Inclusion Criteria:

1. Ages are from 18 to 50;
2. Meeting the criteria of the Diagnostic and Statistical Manual of Mental Disorder (DSM-5) for current unipolar MDD, which is assessed by at least one professional psychiatrist;
3. Han ethnicity;
4. Right handedness;
5. With a score≥17 on the HAMD-1713;
6. With a score≥6 on the BSI14;
7. Without any pharmacotherapy at baseline or maintaining actual pharmacotherapy for at least 2 weeks before the stimulation initiation and during the total stimulation period.

Exclusion Criteria:

1. Assessed through applying the Mini-International Neuropsychiatric Interview (MINI)15 by professional psychiatrists that diagnosed any other current or past psychiatric axis-I disorders (except MDD in the patients);
2. Severe liver and kidney diseases, active endocrine diseases or clinical symptoms. Severe cardiovascular disease, respiratory system disease, haematologic diseases and cancer;
3. Any clinically significant abnormal laboratory examination that may influence the health of participants;
4. A history of any aignificant medical illness such as neurological disorders (such as cerebral trauma, seizure disorder, etc);
5. Known current psychosis as determined by the DSM-5 or a history of a non-mood psychotic disorder;
6. Current alcohol and drug abuse;
7. Pregnancy or lactation;
8. Abnormal scalp such as open wounds;
9. HAMD-17 item 3 (suicide) score=4;
10. Receiving modified electroconvulsive therapy (MECT) or repetitive transcranial magnetic stimulation (rTMS) in the past 1 month;
11. Participation in another clinical trial concurrently or no more than 1 month prior to randomisation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Beck rating scale for suicidal ideation (BSI) | At week 1 and week 2
  Change from Baseline BSI at week 1 and week 2

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Chen, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Lyu D, Wang F, Huang Q, Yang W, Zhang M, Wei Z, Shi S, Kong S, Chen S, He S, Yang V, Fang Y, Douiri A, Hong W. Adjunctive duration-doubled transcranial direct current stimulation for the treatment of depressive patients with suicidal ideation: study protocol for a double-blind, randomized, sham-controlled trial. Trials. 2024 Jan 2;25(1):15. doi: 10.1186/s13063-023-07858-0. PMID 38167178